CLINICAL TRIAL: NCT04417803
Title: Interest of Individual Biomarkers From the Identification of Tumor Genotype in Plasma (ctDNA: Circulating Tumor DNA) by High-throughput Molecular Next Generation Techniques(CAPP Seq, PhAsE Seq, VIRCAPP-seq) in the Diagnosis and Personalized Management of Lymphomas in a Prospective Monocentric Cohort
Brief Title: Interest of Individual Biomarkers From the Identification of Tumor Genotype by High-throughput Molecular Techniques
Acronym: BIOLYMPH2020
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ROSSI 2020
Record Dates: First submitted 2020-05-28; First posted 2020-06-05 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Lymphomas
MeSH Terms: conditions — Lymphoma | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- diffuse large B-cell lymphoma (Other)
  Interventions: Biological: Blood sampling
- follicular lymphoma (Other)
  Interventions: Biological: Blood sampling
- Hodgkin's lymphoma (Other)
  Interventions: Biological: Blood sampling
- mantle cell lymphoma (Other)
  Interventions: Biological: Blood sampling
- T-cell lymphomas (Other)
  Interventions: Biological: Blood sampling

INTERVENTIONS:
Biological: Blood sampling — plasmatic sampling

SUMMARY:
Lymphomas are the most common haemopathic malignancy. The 3 most common types are diffuse large B-cell lymphoma (DLBCL), Hodgkin's lymphoma (HL) and follicular lymphoma (FL). In these three subtypes, the treatment strategy is most often curative. The therapeutic strategy is guided by PET (positron emission tomography), which optimises the risk-benefit balance between the efficacy and toxicity of the treatment and makes it possible to limit the intensity of treatment for good responders and to intensify the treatment of poor responders with a worse prognosis. PET therefore plays a central role in the pre-therapeutic evaluation of the disease and in the assessment of response to treatment. However, other complementary approaches could improve characterization prior to initiating lymphoma t-treatment and individual patient management during treatment and beyond. In DLBCL, it has been shown that the risk of relapse of good and bad responders is decreased by combining the PET response with a reduction in the amount of tumor DNA (ctDNA) in the blood, i.e. the genetic program of lymphoma cells that circulates freely in the blood. This evaluation of ctDNA has been made possible by the development of innovative techniques such as Next Generation Sequencing (NGS). In lymphomas, several approaches have been developed, the most sensitive and promising being CAPP-Seq (CAncer Personalized Profiling by deep Sequencing) developed at Stanford University.

It is therefore useful to study the description of ctDNA in the 3 types of lymphomas and to analyse the progression profiles under treatment by trying to establish the major potential usefulness of these techniques: modifying treatment in case of poor response based on ctDNA +/- and PET, detecting relapses earlier than at present in patients without any other sign of relapse (clinical, blood or PET).

The project presented here aims to build a collection of plasma samples taken before treatment, during treatment and during the first 2 years of follow-up in patients with one of the 3 most frequent types of lymphoma and undergoing curative treatment. The hypothesis is that sequential evaluation of ctDNA could improve the individualized management of future patients based on the results generated by the analyses of patients in this cohort.

Given the progress made in setting up this tool for DLBCL and HL, it is highly appropriate to explore its potential usefulness in other subtypes such as mantle cell lymphoma (MCL) and T-cell lymphoma (TL).

ELIGIBILITY:
Inclusion Criteria:

* Person who has not opposed to their inclusion in the trial
* Confirmation of the diagnosis of one of the lymphomas (DGLBL, LF, classic LH, LT or LCM) according to the WHO 2016 international classification (Smerdlow et al, 2016)
* Patients not currently taking treatment for their haemopathy (or who have received corticosteroid therapy alone within 14 days prior to the 1st sampling, dose limited to 500mg total)
* Patients requiring systemic treatment within 30 days of screening

Exclusion Criteria:

* Person subject to legal protection (curatorship, guardianship)
* Person under partial judicial control
* Pregnant, parturient or breastfeeding woman
* Adult incapable or incapable to express his or her non-opposition
* Minor
* Localized lymphoma treated by surgery and/or localized radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2021-05-17 (Actual); Primary Completion 2046-05 (Estimated); Study Completion 2046-05 (Estimated)

PRIMARY OUTCOMES:
biomarkers | through study completion, an average of 7 years
  identification of individual plasma biomarkers, based on cfDNA (cell-free DNA), by high-throughput sequencing of circulating ctDNA tumor DNA

SECONDARY OUTCOMES:
tumour mutation profile | through study completion, an average of 7 years
  Description of the tumour mutation profile using different molecular biology techniques (CAPP-seq, PHASE-seq, VIRCAPP-seq) by analysing circulating tumour DNA (ctDNA) from cfDNA

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France

IPD SHARING:
Plan to Share IPD: No